CLINICAL TRIAL: NCT07322601
Title: Evaluation of the Supportive Analgesic Effect of Auricular Acupressure After Cesarean Section: A Randomized Clinical Controlled Trial
Brief Title: Supportive Analgesic Effect of Auricular Acupressure (AA) After Cesarean Section (CS)
Acronym: AA-CS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Lê Phương Linh, Medical Doctor, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 3962/DHYD-HDDD
Record Dates: First submitted 2025-12-14; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-10

CONDITIONS: Pain Postoperative; Caesarean Section; Pain
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Acupuncture, Ear; Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to the auricular acupressure group or sham auricular acupressure group in a 1:1 ratio.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auricular Acupressure Group (Experimental): Participants received auricular acupressure using Vaccaria seeds applied to Shenmen [Antitragus-4 (TF4)], Lung [Concha-14 (CO14)], Internal Genitalia [Triangular fossa-2 (TF2)], Pelvis [Triangular fossa-5 (TF5)], Subcortex [Antitragus-4 (AT4)], and Sympathetic [Antihelix-6 (AH6)].
  Interventions: Other: Auricular Acupressure
- Sham Auricular Acupressure Group (Sham Comparator): Participants received identical adhesive patches without seeds applied to the same auricular points.
  Interventions: Other: Sham Auricular Acupressure Group

INTERVENTIONS:
Other: Auricular Acupressure — In the Auricular Acupressure group, participants received auricular acupressure using vaccaria seeds applied to the following points on both ears: Ear Shenmen (TF4), Lung (CO14), Internal Genitalia (TF2), Pelvis (TF5), Subcortex (AT4), and Sympathetic (AH6), in addition to standard postoperative care.
  Each participant received a single treatment session within 5 hours after cesarean section, once transferred to the Obstetrics Department. Seeds were retained for 2 days. All acupuncture procedures were performed by licensed traditional medicine physicians who had been trained and standardized before the study.
  Other Names: Auricular Acupuncture; Acupuncture
  Arms: Auricular Acupressure Group
Other: Sham Auricular Acupressure Group — In the Sham Auricular Acupressure Group, participants received adhesive patches without seeds, identical in size and appearance to the Auricular Acupressure Group patches, applied to the same auricular points. Both groups received standard postoperative care.
  Other Names: Sham Acupuncture; Sham Auricular Acupuncture
  Arms: Sham Auricular Acupressure Group

SUMMARY:
Introduction:

Severe acute pain after cesarean section is an independent risk factor for the development of chronic pain and increases the risk of postpartum depression threefold. Pain also reduces the mother's ability to breastfeed and care for her child. This study aimed to evaluate the supportive effectiveness of auricular acupressure in reducing incision pain and uterine contraction pain in women undergoing cesarean section, compared with sham auricular acupressure.

Methods:

A randomized, controlled, single-blind clinical trial was conducted in seventy women undergoing cesarean section, randomly allocated (1:1) to an auricular acupressure or sham group. The study group received vaccaria seeds, and the sham group received non-vaccaria patches on both ears. Both groups were treated at the Shenmen, Lung, Internal Genitalia, Pelvis, Subcortex, and Sympathetic points. Pain was assessed using the Visual Analog Scale (VAS), and diclofenac consumption was recorded over the first 48 hours postpartum.

DETAILED DESCRIPTION:
Participants are instructed to apply pressure to the patches three times daily (morning, noon, and evening). Supplemental acupressure is also performed whenever the participant feels pain, with the goal of achieving the 'De-qi' sensation (a feeling of soreness or tingling). All patches are maintained for 48 hours. Postoperative analgesia follows a standardized hospital protocol, with diclofenac administered as rescue medication.

Safety monitoring is strictly implemented throughout the study. If participants experience symptoms such as headache, dizziness, or syncope following the application of auricular patches, they will be managed according to standardized acupuncture safety protocols. Participants will be withdrawn from the study if they develop adverse reactions, including local allergic reactions at the patch site, persistent local pain, or severe dizziness.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years of age
* Gestational age ≥ 37 weeks
* Alert and cooperative with the treating physicians
* Able to understand and use the Visual Analog Scale (VAS)
* Preoperative American Society of Anesthesiologists (ASA) Physical Status Classification System I-II
* Anesthesia: spinal anesthesia;
* Pfannenstiel suprapubic transverse incision
* Infant 5-minute Appearance, Pulse, Grimace, Activity, Respiration score (Apgar score) > 7
* Cesarean operative time ≤ 60 minutes
* Singleton pregnancy
* Voluntary agreement to participate.

Exclusion Criteria:

* Contraindication to diclofenac
* Surgical complications, including hysterectomy and postpartum hemorrhage (> 1000 ml)
* History of acupuncture syncope
* Preoperative chronic pain and/or regular preoperative use of analgesics
* Addiction to or dependence on opioids or alcohol
* Diabetes mellitus or HIV infection
* Prior Auricular acupressure
* Skin lesions of the auricle
* Surgical wound infection

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 70 (Actual)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Pain relief effectiveness was assessed using the Visual Analog Scale (VAS) for pain intensity at rest, during movement and for uterine contractions at 12, 24, and 48 hours after cesarean section. | 12, 24, 48 hours postoperative
  Pain relief effectiveness was assessed using the Visual Analog Scale (VAS) for pain intensity at rest, during movement and for uterine contractions at 12, 24, and 48 hours after cesarean section. The Visual Analog Scale (VAS) consists of a line where respondents are asked to mark their level of pain. The left-most point (zero) represents no pain and the right-most point (10) represents extreme pain. The higher the score, the more severe the pain.
VAS scores for pain intensity at rest, pain intensity on movement, and uterine contraction pain | From enrollment to the end of treatment at 48 hours
  Pain relief effectiveness was assessed using the Visual Analog Scale (VAS) for pain intensity at rest, during movement and for uterine contractions at 12, 24, and 48 hours after cesarean section. The Visual Analog Scale (VAS) consists of a line where respondents are asked to mark their level of pain. The left-most point (0) represents 'no pain,' while the right-most point (10) represents 'extreme pain.' The higher the score, the more severe the pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ly, PhD, Study Chair — University of Medicine and Pharmacy at Ho Chi Minh City
Locations (1):
- Le Van Thinh Hospital, Ho Chi Minh City, Binh Trung Ward, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
The type of data set or supporting information being shared. Options include: study protocol, statistical analysis plan, informed consent form, clinical study report, analytic code.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 3 years after the publication of results
Access Criteria: Data will be made available to qualified researchers for the purpose of valid scientific research. To gain access, investigators must submit a formal research proposal and a statistically sound analysis plan to the Principal Investigator. All requests will be reviewed by the study's investigators and the Institutional Ethics Committee. Upon approval, requestors will be required to sign a Data Use Agreement (DUA) to ensure participant confidentiality. The shared data will be de-identified and may include the study protocol and statistical analysis plan.